CLINICAL TRIAL: NCT00660166
Title: HLA Class I Haplotype Mismatched Natural Killer Cell Infusions After Autologous Stem Cell Transplant for Hematological Malignancies
Brief Title: Human Leukocyte Antigen (HLA) Class I Haplotype Mismatched Natural Killer Cell Infusions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Allogeneic NKCell post ABMT
Record Dates: First submitted 2008-04-11; First posted 2008-04-17 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Lymphoma; Myeloma; Leukemia
Keywords: Natural killer cells; autologous stem cell transplant; immunotherapy
MeSH Terms: conditions — Lymphoma; Neoplasms, Plasma Cell; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: NK-Cell Infusion

INTERVENTIONS:
Biological: NK-Cell Infusion — The infusion of natural killer (NK) cells will be performed in the Infusion Center at New England Medical Center. The NK cells will be given to the subject intravenously (into a vein). In addition, a balanced salt solution will be infused beginning about two hours prior to and continuing for two hours after the infusion of NK cells to keep the fluid level in the body well balanced. The subject will also receive Benadryl by injection 15-30 minutes prior to infusion to counteract and prevent any unwanted allergic side effects. The subject will be observed for any side effects during this time. If the subject feels well, he/she can go home. However, there may be a requirement to keep him/her overnight.

SUMMARY:
The purpose of this research study is to examine the safety of infusing escalated doses of allogeneic (from a relative of the patient), enriched natural killer (NK) cells after autologous (from the patient) stem cell transplantation. The hypothesis is that the infusion of these NK cells early after an autologous stem cell transplant will help to eliminate and eradicate any residual cancerous cells that remain in the body and may have survived the chemotherapy or radiation.

DETAILED DESCRIPTION:
Natural killer cells are blood cells that are responsible for eliminating cancer cells especially when there are only a few. It has been shown that NK cells coming from a "mismatched" person (a relative) have a better chance than the patient's own NK cells to recognize and kill cancer cells. These cells will be collected from the blood of a parent, child or sibling and after preparation in the laboratory, will be given to the patient early after an autologous stem cell transplantation like a blood or platelet transfusion. A person who has been diagnosed with a blood tumor and received an autologous stem cell transplant has the chance of his/her cancer coming back. This study uses NK cells obtained from a relative to prevent disease recurrence by potentially eliminating and eradicating any residual cancerous cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone an autologous stem cell transplant for the following diseases:

  * Acute Myeloid Leukemia
  * Non-Hodgkin's Lymphoma
  * Hodgkin's Disease
  * Multiple Myeloma
* Age 13 - 70 years old
* Able to give informed consent
* Hepatic and renal function: bilirubin less than or equal to 2x normal limits, AST and ALT less than or equal to 2x normal limits, serum creatinine less than or equal to 1.5x normal
* ECOG Performance Status less than or equal to 1 (at planned time of transplantation)
* Patients with no active infection

Exclusion Criteria:

* Patients who have not recovered sufficiently from the side effects of the autologous transplant (i.e. have > grade 2 toxicity in any organ system)
* Patients who have insufficient engraftment parameters according to the following criteria: WBC < 2,500 /mm3 and platelets < 50,000/mm3
* Radiation therapy, chemotherapy, or immunotherapy beginning one week before NK-cell infusion and lasting 2 weeks after NK-cell infusion.
* Intrinsic impaired organ function (as stated above).
* Physical or psychiatric conditions that in the estimation of the PI or designee place the patient at high-risk of toxicity or non-compliance.
* Uncontrolled, life-threatening infections at the time of infusion.
* Concurrent treatment with corticosteroids and/or other immuno-suppressive drugs.

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
An evaluation of general safety will be undertaken: · Number of systemic clinical and biological adverse events occurring during the study. · Number of patients who prematurely discontinued study treatment for reasons linked to the general safety. | 58 days post infusion of allogeneic NK-cells

SECONDARY OUTCOMES:
Duration of donor NK cells in the recipient's blood | 58 days post infusion of allogeneic NK-cells
Patient survival at 100 days and at one year post treatment (all cause mortality) | 100 days and one year post treatment
Occurrence of new cancer during the first year post infusion of allogeneic NK-cells | One year post infusion of allogeneic NK-cells
Documented systemic infections during the first 30 days post infusion of allogeneic NK-cells. | 30 days post infusion of allogeneic NK-cells
Occurrence of other possible NK-infusions related complications such as,fever, capillary leak syndrome and/or allergic reaction. | 58 days post infusion of allogeneic NK-cells

CONTACTS AND LOCATIONS:
Overall Officials: Hans Klingemann, MD, PhD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Klingemann H, Boissel L. Targeted cellular therapy with natural killer cells. Horm Metab Res. 2008 Feb;40(2):122-5. doi: 10.1055/s-2007-1004576. PMID 18283630
- [Result] Klingemann HG. Natural killer cell-based immunotherapeutic strategies. Cytotherapy. 2005;7(1):16-22. doi: 10.1080/14653240510018000. PMID 16040380